CLINICAL TRIAL: NCT03418181
Title: Does Incremental Initiation of Haemodialysis Preserve Native Kidney Function? A Multicentre Feasibility Randomised Controlled Trial
Brief Title: Does Incremental Initiation of Haemodialysis Preserve Native Kidney Function?
Acronym: IncrementalHD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: East and North Hertfordshire NHS Trust (Other Government)
Collaborators: University of Hertfordshire (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RD2017-21
Record Dates: First submitted 2017-09-20; First posted 2018-02-01 (Actual); Last update posted 2018-02-01 (Actual); Status verified 2018-01

CONDITIONS: Kidney Failure; Dialysis
Keywords: Residual Kidney Function; Haemodialysis; Preserve Residual Kidney Function
MeSH Terms: conditions — Renal Insufficiency

STUDY DESIGN:
Intervention Model Description: The participants will be randomly allocated to 2 groups:
  1. Thrice weekly dialysis (control arm)
  2. Incremental dialysis - Twice weekly dialysis to start with and slowly increasing the duration and frequency of dialysis to thrice weekly depending on their native kidney function.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Haemodialysis (Other): Thrice weekly dialysis (control arm) - dialysis dose will not be adjusted according to Residual Kidney Function and subjects will be dialysed initially for 3.5-4 hours thrice weekly to ensure a target minimum eKt/V of 1.2.
  Interventions: Procedure: Standard Haemodialysis
- Incremental dialysis (Experimental): Twice weekly dialysis - dialysis dose will be adjusted according to Residual Kidney Function.
  Patients will commence dialysis for 3.5-4 hours twice weekly and have residual renal urea clearance formally measured by interdialytic urine collection at the end of the week following dialysis initiation. Subsequent to this, dialysis dose will be adjusted.
  Interventions: Procedure: Incremental dialysis

INTERVENTIONS:
Procedure: Standard Haemodialysis — Thrice weekly dialysis.
  Arms: Standard Haemodialysis
Procedure: Incremental dialysis — Individualised dialysis dose according to native kidney function.
  Arms: Incremental dialysis

SUMMARY:
Patients who start haemodialysis usually retain some natural kidney function for months or years after starting dialysis. Even a small amount of this natural kidney function can be helpful in reducing the need for dietary and fluid restriction. There is also good evidence that retaining a small amount of natural kidney function may provide a survival benefit for patients on dialysis.

Most patients who commence haemodialysis start three times per week for 3.5-4 hours per session, irrespective of the amount of natural kidney function they may have. An alternative approach used in some kidney units is to take account of the natural kidney function in prescribing the amount of dialysis. This may allow patients to start treatment needing to spend less time on dialysis or even to start just twice weekly. The amount of dialysis can be adjusted over time as natural kidney function declines. This is called "incremental haemodialysis". Both of these approaches are considered to be standard care although it is not known which approach is more beneficial to patients.

There are some suggestions that the frequency of dialysis may influence the rate of decline of natural kidney function but this need to be tested in a large randomised study. To inform the design of such a study, a smaller scale feasibility study is required.

We intend to randomise fifty new starters on haemodialysis with adequate natural kidney function into two groups - a group who will have dialysis prescribed in the standard fashion - three times weekly for 3.5-4 hours per session or a group who will have an incremental start beginning with twice weekly treatment. We will investigate how many patients have sufficient natural kidney function to be eligible, whether patients are willing to participate and continue in the study, compare the rate of loss of kidney function between groups, and ascertain whether this individualised dialysis approach is less intrusive to patients. The results will be used to design a larger definitive study.

DETAILED DESCRIPTION:
This study is feasibility randomised controlled trial.

50 patients who have newly started on haemodialysis will be recruited into the study from 4 UK centres.

Eligible patients will be approached prior to initiation of dialysis or after starting dialysis. The details of the study will be explained to them and a Patient Information sheet will be provided. Interested participants will be invited to the study and a written consent will be obtained.

The participants will be randomly allocated to 2 groups.

1. Thrice weekly dialysis (control arm)
2. Incremental dialysis - Twice weekly dialysis to start with and slowly increasing the duration and frequency of dialysis to thrice weekly depending on their native kidney function.

All participants will be monitored at least once monthly by performing dialysis related blood tests, urine tests, clinical evaluation, medications, weight, dialysis adequacy, adverse events.

Questionnaire involving quality of life, mood, illness intrusiveness, functional status, cognitive function will also be performed.

Participants will be recruited in the first year and all participants will be followed up for 12 months. All participants may withdraw at any time without any change in their dialysis care.

To ensure independence, the University of Hertfordshire will perform randomisation, and assist with data monitoring and data analysis.

A 6 month rate of loss of native kidney function between the 2 groups will be analysed.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Advanced renal failure due to underlying primary kidney disease and established as a new starter on haemodialysis within the previous 3 months
* Residual Kidney Function likely to permit twice weekly dialysis as defined by interdialytic urea clearance ≥3ml/min/1.73m2 BSA measured routinely as part of standard care
* Sufficient understanding of the study procedures and requirements including capacity for explicit agreement to be randomised to standard or incremental HD regimens

Exclusion Criteria:

* Planned organ transplantation and already on another interventional trial within 3 months from study screening
* Anticipated requirement for high-volume ultrafiltration on dialysis (e.g. subjects with daily enteral or parenteral nutrition)
* Blood-borne virus positivity
* Subjects unable to comply with requirement for monthly interdialytic urine collection.
* Pregnancy
* Prognosis <12 months as judged by PI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-01-08 (Actual); Primary Completion 2019-01-02 (Estimated); Study Completion 2019-03-02 (Estimated)

PRIMARY OUTCOMES:
Recruitability | 12 months
  Number of patients potentially eligible for screening during the study period
Recruitability | 12 months
  Proportion of screened patients who fulfil study criteria.
Recruitability | 12 months
  Proportion of patients approached who agree to participate in the study.
Retainability | 12 months
  Proportion of patients randomised who withdraw from the study and the reasons for their withdrawal.
Protocol Adherence | 12 months
  Proportion of patients who adhere to protocol dialysis frequency.
Incidence of hospital admissions due to hyperkalemia, fluid overload, lower respiratory tract infection [Safety of the study] | 12 months
  Frequency of hospital admission due to hyperkalemia and fluid overload, and lower respiratory tract infection (LRTI).
Effect size | 6 months after randomisation
  Rate of change (mean) of RKF in the first 6 months after randomisation.
Dialysis dose | 6 months after randomisation
  Dialysis dose measured by eKT/V
Residual kidney function | 6 months after randomisation
  Residual kidney function measured by eKT/V

SECONDARY OUTCOMES:
Quality of life | 12 months
  Assessed using EQ-5D-5L questionnaire.
Depression | 12 months
  Assessed using PHQ-9 questionnaire.
Illness intrusiveness | 12 months
  Assessed using Illness intrusiveness rating scale.
Changes in cognitive function | 12 months
  Assessed by MOCA tool.
Functional status | 12 months
  Assessed by Clinical Frailty Score (CFS).
Incidence of vascular access failures [Safety] | 12 months
  Frequency of vascular access failures and interventions.
Major Adverse Cardiac Events | 12 months
  Assessed by recording of the frequency of the events.
Survival | 12 months
  Measured by all-cause mortality

CONTACTS AND LOCATIONS:
Overall Officials: Dr Enric Vilar, Principal Investigator — East and North Hertfordshire NHS Trust
Locations (1):
- East and North Hertfordshire NHS Trust (incorporating Mount Vernon Cancer Centre), Stevenage, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Identifiable personal data will not be published. Study results will be reported to the British Renal Society Conference and published in peer-reviewed journal, presented in conferences (up to 5 years).

REFERENCES:
- [Derived] Kaja Kamal RM, Farrington K, Wellsted D, Sridharan S, Alchi B, Burton J, Davenport A, Vilar E. Impact of incremental versus conventional initiation of haemodialysis on residual kidney function: study protocol for a multicentre feasibility randomised controlled trial. BMJ Open. 2020 Aug 13;10(8):e035919. doi: 10.1136/bmjopen-2019-035919. PMID 32792431